CLINICAL TRIAL: NCT01749748
Title: The Study of Breast MRI Screening and Proton Magnetic Resonance Spectroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Hospital, physician, clinical assistant professor, principal investigator of Department of Medical Imaging, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200806009R
Record Dates: First submitted 2012-11-17; First posted 2012-12-17 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Breast Diseases
Keywords: Breast diseases; magnetic resonance spectroscopy
MeSH Terms: conditions — Breast Diseases | interventions — Proton Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- proton magnetic resonance spectroscopy (Other): proton magnetic resonance spectroscopy for asymptomatic women breasts.
  Interventions: Procedure: proton magnetic resonance spectroscopy

INTERVENTIONS:
Procedure: proton magnetic resonance spectroscopy — proton magnetic resonance spectroscopy was performed for the normal breast to evaluate the chemical composition of breast
  Other Names: proton MRS

SUMMARY:
To delineate if the chemical composition (lipid and water) in the presumably normal breast of the high risk women is different from those of the low risk group.

DETAILED DESCRIPTION:
The researchers would like to investigate and compare the chemical composition in the normal breast between high risk women and general population.

ELIGIBILITY:
Inclusion Criteria:

* Women without breast symptoms (without family history of breast cancer; or with at least first-degree relative of breast cancer) with negative mammography and ultrasound result in recent 3 months or contralateral normal breasts from women with newly diagnosed unilateral breast cancer
* 25-75 years old.

Exclusion Criteria:

* renal function impairment
* past history of anaphylactoid reaction to MRI contrast media (Gd-DTPA)
* pregnant or lactating women
* medication of HRT or oral pills in recent 6 months
* past history of surgery of the breast (either side)
* past history of breast cancer
* with breast implant or silicone injection
* past history of cardiac surgery, mechanical valve replacement, aneurismal clip, endotracheal tube or tracheostomy tube, any metallic implants.

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2008-07; Primary Completion 2015-08 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
comparison of lipid water composition and ratio of the normal breasts in women of high risk group and low risk group. | up to 5 years ( July 2008 to June 2013)
  This is a cross sectional study. And we just assess the chemical composition of normal breasts of women at a given time point, since the participants only received one time of study.

SECONDARY OUTCOMES:
to investigate the association between breast density and lipid water ratio of normal breasts | up to 5 years (July 2008 to June 2013)
  to investigate whether there is association of breast density and chemical composition of normal breast on proton magnetic resonance spectroscopy.
to investigate the association between menopausal status and lipid water ratio of normal breasts | up to 5 years ( July 2008 to June 2013)
  to investigate whether there is association of menopausal status and chemical composition of normal breast on proton magnetic resonance spectroscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Jane Wang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan